CLINICAL TRIAL: NCT01633333
Title: Water Exchange Versus Carbon Dioxide Insufflation to Improve Colonoscopy Screening - a Randomized Controlled Trial
Brief Title: Water Exchange Versus Carbon Dioxide for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WMCO2_KG
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Colorectal Cancer; Colorectal Adenomas; Colorectal Polyps; Pain
Keywords: Colonoscopy; Colorectal cancer; Colorectal adenomas; Pain
MeSH Terms: conditions — Colorectal Neoplasms; Pain | interventions — Carbon Dioxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water exchange (Experimental): Colonoscopy with water exchange as the sole modality to reach the cecum. Carbon dioxide can be used in case of intubation failure with the test method.
  Interventions: Other: Water exchange colonoscopy
- Carbon dioxide insufflation (Active Comparator): Carbon dioxide insufflation will be used in standard fashion to reach the cecum.
  Interventions: Other: Carbon dioxide insufflation

INTERVENTIONS:
Other: Water exchange colonoscopy — Water is infused and suctioned in a systematic fashion to obtain luminal view and for cleansing of the colon to facilitate colonoscope insertion. The carbon dioxide pump is turned off, only to be turned on during withdrawal from the cecum.
  Other Names: Water exchange
  Arms: Water exchange
Other: Carbon dioxide insufflation — Carbon dioxide insufflation to obtain luminal view to facilitate colonoscope insertion, considered to be standard procedure.
  Other Names: Carbon dioxide
  Arms: Carbon dioxide insufflation

SUMMARY:
Colonoscopy is commonly used in screening for colorectal cancer. A refined technique of colonoscopy involving the use of water as the sole modality to aid colonoscope insertion, water exchange, has been described in recent research papers to decrease patient discomfort and pain, and to reduce the need for sedation during colonoscopy when compared with standard air insufflation. Carbon dioxide insufflation has been described to decrease patient discomfort after colonoscopy. No randomized trial has so far compared the use of water exchange to carbon dioxide insufflation. Our hypothesis is that water exchange inflicts less discomfort to patients undergoing colonoscopy than carbon dioxide insufflation. Patients undergoing screening colonoscopy in two centers in Norway, one center in Poland and one center in The Netherlands will be enrolled and randomized to examination of either of the two methods.

DETAILED DESCRIPTION:
Single blinded randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for screening or polyp surveillance colonoscopy
* Patients accepting sedation on demand

Exclusion Criteria:

* Demand for sedation/analgesia before the start of the procedure
* Previous partial or total colonic resection
* Pregnancy
* Unwilling/unable to provide informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain during colonoscopy | 1 hour
  Patients will be asked by a blinded assistant immediately after colonoscopy to score pain during the procedure.

SECONDARY OUTCOMES:
Pain during colonoscopy | 30 minutes
  Patients will be asked to report pain during colonoscopy to an unblinded study assistant.
Cecal intubation rate | 1 hour
  Cecal intubation rate is defined as successful completion of colonoscopy insertion. This will be analyzed on an intention-to-treat basis according to group allocation.
Cecal intubation time | 1 hour
  The time taken to complete insertion of the colonoscope.
Adenoma detection rate | 1 hour
  Detection of adenomas during each colonoscopy procedure
Polyp detection rate | 1 hour
  Detection of any colonic polyp, irrespective of histologic type, during each procedure.
Dose of medication | 1 hour
  Dose of sedative and analgesic medication needed to complete the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil K Garborg, MD, Principal Investigator — Sorlandet Hospital HF Kristiansand, Norway
Locations (3):
- Norway (2):
  - Sorlandet Hospital, Arendal
  - Sorlandet Hospital, Kristiansand
- The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland

REFERENCES:
- [Background] Denberg TD, Melhado TV, Coombes JM, Beaty BL, Berman K, Byers TE, Marcus AC, Steiner JF, Ahnen DJ. Predictors of nonadherence to screening colonoscopy. J Gen Intern Med. 2005 Nov;20(11):989-95. doi: 10.1111/j.1525-1497.2005.00164.x. PMID 16307622
- [Background] Khalid-de Bakker CA, Jonkers DM, Hameeteman W, de Ridder RJ, Masclee AA, Stockbrugger RW. Cardiopulmonary events during primary colonoscopy screening in an average risk population. Neth J Med. 2011 Apr;69(4):186-91. PMID 21527807
- [Background] Jonas DE, Russell LB, Sandler RS, Chou J, Pignone M. Patient time requirements for screening colonoscopy. Am J Gastroenterol. 2007 Nov;102(11):2401-10. doi: 10.1111/j.1572-0241.2007.01387.x. Epub 2007 Jun 29. PMID 17608779
- [Background] Leung FW, Leung JW, Mann SK, Friedland S, Ramirez FC. The water method significantly enhances patient-centered outcomes in sedated and unsedated colonoscopy. Endoscopy. 2011 Sep;43(9):816-21. doi: 10.1055/s-0030-1256407. Epub 2011 May 24. PMID 21611947
- [Background] Ramirez FC, Leung FW. A head-to-head comparison of the water vs. air method in patients undergoing screening colonoscopy. J Interv Gastroenterol. 2011 Jul;1(3):130-135. doi: 10.4161/jig.1.3.18512. Epub 2011 Jul 1. PMID 22163084
- [Background] Leung FW, Leung JW, Siao-Salera RM, Mann SK, Jackson G. The water method significantly enhances detection of diminutive lesions (adenoma and hyperplastic polyp combined) in the proximal colon in screening colonoscopy - data derived from two RCT in US veterans. J Interv Gastroenterol. 2011 Apr;1(2):48-52. doi: 10.4161/jig.1.2.16826. PMID 21776425
- [Background] Leung F, Harker J, Leung J, Siao-Salera R, Mann S, Ramirez F, Friedland S, Amato A, Radaelli F, Paggi S, Terruzzi V, Hsieh Y. Removal of infused water predominantly during insertion (water exchange) is consistently associated with a greater reduction of pain score - review of randomized controlled trials (RCTs) of water method colonoscopy. J Interv Gastroenterol. 2011 Jul;1(3):114-120. doi: 10.4161/jig.1.3.18510. Epub 2011 Jul 1. PMID 22163081
- [Background] Leung F, Harker J, Leung J, Siao-Salera R, Mann S, Ramirez F, Friedland S, Amato A, Radaelli F, Paggi S, Terruzzi V, Hsieh Y. Removal of infused water predominantly during insertion (water exchange) is consistently associated with an increase in adenoma detection rate - review of data in randomized controlled trials (RCTs) of water-related methods. J Interv Gastroenterol. 2011 Jul;1(3):121-126. doi: 10.4161/jig.1.3.18517. Epub 2011 Jul 1. PMID 22163082
- [Background] Stevenson GW, Wilson JA, Wilkinson J, Norman G, Goodacre RL. Pain following colonoscopy: elimination with carbon dioxide. Gastrointest Endosc. 1992 Sep-Oct;38(5):564-7. doi: 10.1016/s0016-5107(92)70517-3. PMID 1397911
- [Background] Bretthauer M, Thiis-Evensen E, Huppertz-Hauss G, Gisselsson L, Grotmol T, Skovlund E, Hoff G. NORCCAP (Norwegian colorectal cancer prevention): a randomised trial to assess the safety and efficacy of carbon dioxide versus air insufflation in colonoscopy. Gut. 2002 May;50(5):604-7. doi: 10.1136/gut.50.5.604. PMID 11950803
- [Background] Sumanac K, Zealley I, Fox BM, Rawlinson J, Salena B, Marshall JK, Stevenson GW, Hunt RH. Minimizing postcolonoscopy abdominal pain by using CO(2) insufflation: a prospective, randomized, double blind, controlled trial evaluating a new commercially available CO(2) delivery system. Gastrointest Endosc. 2002 Aug;56(2):190-4. doi: 10.1016/s0016-5107(02)70176-4. PMID 12145595
- [Background] Church J, Delaney C. Randomized, controlled trial of carbon dioxide insufflation during colonoscopy. Dis Colon Rectum. 2003 Mar;46(3):322-6. doi: 10.1007/s10350-004-6549-6. PMID 12626906
- [Background] Wong JC, Yau KK, Cheung HY, Wong DC, Chung CC, Li MK. Towards painless colonoscopy: a randomized controlled trial on carbon dioxide-insufflating colonoscopy. ANZ J Surg. 2008 Oct;78(10):871-4. doi: 10.1111/j.1445-2197.2008.04683.x. PMID 18959640
- [Background] Uraoka T, Kato J, Kuriyama M, Hori K, Ishikawa S, Harada K, Takemoto K, Hiraoka S, Fujita H, Horii J, Saito Y, Yamamoto K. CO(2) insufflation for potentially difficult colonoscopies: efficacy when used by less experienced colonoscopists. World J Gastroenterol. 2009 Nov 7;15(41):5186-92. doi: 10.3748/wjg.15.5186. PMID 19891018
- [Background] Riss S, Akan B, Mikola B, Rieder E, Karner-Hanusch J, Dirlea D, Mittlbock M, Weiser FA. CO2 insufflation during colonoscopy decreases post-interventional pain in deeply sedated patients: a randomized controlled trial. Wien Klin Wochenschr. 2009;121(13-14):464-8. doi: 10.1007/s00508-009-1202-y. PMID 19657610
- [Background] Geyer M, Guller U, Beglinger C. Carbon dioxide insufflation in routine colonoscopy is safe and more comfortable: results of a randomized controlled double-blinded trial. Diagn Ther Endosc. 2011;2011:378906. doi: 10.1155/2011/378906. Epub 2011 Jun 15. PMID 21747649
- [Background] Leung FW, Leung JW, Mann SK, Friedland S, Ramirez FC, Olafsson S. DDW 2011 cutting edge colonoscopy techniques - state of the art lecture master class - warm water infusion/CO(2) insufflation for colonoscopy. J Interv Gastroenterol. 2011 Apr;1(2):78-82. doi: 10.4161/jig.1.2.16830. PMID 21776430
- [Background] Hoff G, Bretthauer M, Huppertz-Hauss G, Kittang E, Stallemo A, Hoie O, Dahler S, Nyhus S, Halvorsen FA, Pallenschat J, Vetvik K, Kristian Sandvei P, Friestad J, Pytte R, Coll P. The Norwegian Gastronet project: Continuous quality improvement of colonoscopy in 14 Norwegian centres. Scand J Gastroenterol. 2006 Apr;41(4):481-7. doi: 10.1080/00365520500265208. PMID 16635918
- [Derived] Garborg K, Kaminski MF, Lindenburger W, Wiig H, Hasund A, Wronska E, Bie RB, Kleist B, Lovdal L, Holme O, Kalager M, Hoff G, Bretthauer M. Water exchange versus carbon dioxide insufflation in unsedated colonoscopy: a multicenter randomized controlled trial. Endoscopy. 2015 Mar;47(3):192-9. doi: 10.1055/s-0034-1390795. Epub 2014 Nov 20. PMID 25412093